CLINICAL TRIAL: NCT02761772
Title: Prospective Early Pregnancy Cohort and Preimplantation Factor: Factors Related to Successful Implantation, Risk of Miscarriage and Recurrent Pregnancy Loss in the First Trimester
Brief Title: Early Pregnancy Cohort and Preimplantation Factor
Acronym: PEP-cohort
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Yale University (Other); BioIncept LLC (Industry)
Responsible Party: Principal Investigator, Jesper Friis Petersen, M.D., PhD student, Nordsjaellands Hospital
Other Study IDs: PEP-PIF-2016
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Luteal Phase; Biomarkers; Abortion, Spontaneous; Abortion, Habitual; Pregnancy
Keywords: Preimplantation Factor
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PEP-A: See detailed description
- PEP-S: See detailed description

SUMMARY:
Miscarriage is a common event associated with severe psychological and social morbidity, further tormenting in women suffering recurrent pregnancy loss (RPL) by at least three consecutive losses.

Ultrasonography and biomarkers have yet to precisely predict viability in pregnancies with symptoms of threatening miscarriage.

A novel biomarker Preimplantation Factor (PIF) derived by the developing embryo might be the key factor for this prediction ameliorating the implantation process by promoting a favorable local immune system in the uterus.

The investigators aim to establish a prospective early pregnancy cohort (PEP-cohort) that includes women throughout the first trimester by both assisted reproductive technology (ART) and spontaneous conceptions. By a combination of consecutive ultrasonographys and blood samples of known predictors of implantation PIF as a predictor of viability will be evaluated.

These data are finally compared to the same data in a retrospective cohort of RPL patients emphasizing the role of PIF.

All collected data will be stored in a Research Biobank for the current studies outlined as well as potential future studies of reproductive medicine in the first trimester.

DETAILED DESCRIPTION:
The investigators aim to evaluate Preimplantation Factor (PIF) throughout the first trimester we need to employ two settings of recruitment.

Early part:

The PEP in ART (PEP-A) will enroll participants referred for fertility treatment at Rigshospitalet and North Zealand Hospital. Participants all have cryopreserved embryos suitable for frozen embryo transfer in a natural menstrual cycle. No type of ovulation trigger will be employed, as the LH peak is monitored via home urine-LH test.

For a thorough examination of the luteal phase, participants are recalled for blood samples on day 7, 11, 14 and 16 after positive urine-LH test. Hereafter positive serum human chorionic gonadotropin (hCG) denotes a pregnancy and these participants are offered to continue in the later part of the PEP-cohort.

Late part:

PEP in Spontaneous conceptions (PEP-S) represents the sampling of expected normal pregnancies from the local community. Enrolled at the time of the first positive pregnancy test, participants are expected to be included from approximately 5 weeks of gestation. Hereafter participants are recalled every two weeks for blood sampling and transvaginal ultrasonographys of endometrial thickness until a gestational sac and yolk sac are visible for mean sac diameter measuring and eventually the crown-rump-length.

Research biobank All collected data: questionnaires of medical history before enrollment, ultrasonographys and blood samples of progesterone, 17-OH-progesterone, estradiol, alpha-feto-protein (AFP), pregnancy associated placental protein A (PAPP-A), hCG and PIF are stored in a research biobank.

ELIGIBILITY:
PEP-A

Inclusion Criteria:

1. Women in ART treatment by natural cycle frozen embryo transfer only monitored by urine LH.
2. Age above 18 years.
3. Ability to understand read and write Danish for the informed consent.
4. Planned delivery at the hospitals involved in the project.

Exclusion Criteria:

1. Abnormal uterine anatomy or function already known or estimated at first transvaginal ultrasonography.
2. History of recurrent pregnancy loss.
3. Ongoing or former (at least 12 months of no use) narcotics or alcohol abuse (above 14 units of alcohol per week).
4. Contraindication for pregnancy.

PEP-S

Inclusion Criteria:

1. Spontaneous pregnancy in women above 18 years of age.
2. Gestational age of singleton pregnancy below full eight weeks by first transvaginal ultrasound.
3. Ability to understand read and write Danish for the informed consent.
4. Planned delivery at the hospitals involved in the project.

Exclusion Criteria:

1. All types of ART treatment in the actual pregnancy.
2. Abnormal uterine anatomy or function already known or estimated at first transvaginal ultrasonography.
3. History of recurrent pregnancy loss.
4. Ongoing or former (at least 12 months of no use) narcotics or alcohol abuse (above 14 units of alcohol per week).
5. Contraindication for pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PEP-A: Women in ART treatment by natural cycles of frozen embryo transfer at North Zealand Hospital and Rigshospitalet.
  PEP-S: Women with a positive pregnancy test by spontaneous conception, prior to eight weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
PIF in PEP-A | During 2018
  Serum PIF by gestational age in the luteal phase
Prediction model for the risk of spontaneous abortion | During 2018
  The ability of serum PIF to predict viability of natural pregnancies with and without other biomarkers, ultrasonographys and medical history data.
PIF and recurrent pregnancy loss (RPL) | Late 2018
  Serum PIF levels in a unique retrospective cohort of RPL patients

SECONDARY OUTCOMES:
Hormonal development in the luteal phase | During 2018
  Descriptive overview of natural hormones in the luteal phase and their ability to predict pregnancy and live birth rates

OTHER OUTCOMES:
Research biobank for future use | During 2017
  Establishment of a robust research biobank for future studies in blood derived conditions in the first trimester of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Jesper F Petersen, M. D., Principal Investigator — Nordsjaellands Hospital

IPD SHARING:
Plan to Share IPD: Yes
Following collection, data are planned to be shared within a global archive.

REFERENCES:
- [Derived] Petersen JF, Friis-Hansen LJ, Bryndorf T, Jensen AK, Andersen AN, Lokkegaard E. A Novel Approach to Predicting Early Pregnancy Outcomes Dynamically in a Prospective Cohort Using Repeated Ultrasound and Serum Biomarkers. Reprod Sci. 2023 Dec;30(12):3597-3609. doi: 10.1007/s43032-023-01323-8. Epub 2023 Aug 28. PMID 37640889